CLINICAL TRIAL: NCT06942221
Title: Digital Solutions in Heart Therapy (DIGNITY) - a Randomized Controlled Trial Using Telemedicine for Heart Failure Treatment
Brief Title: Digital Solutions in Heart Therapy (DIGNITY)
Acronym: DIGNITY - HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02601; am24Zhou2
Record Dates: First submitted 2025-01-30; First posted 2025-04-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: guideline-directed medical therapy; telemedicine
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine guided care group (Experimental): Patients will be instructed to response to questions using the App daily. The parameters and questionnaires will be evaluated by the Telemedicine team, and participants will be contacted via phone 1 week after discharge and subsequently every 7-10 days to discuss the up-titration of the HF medications.
  Interventions: Other: guideline-directed medical therapy
- usual care group (Active Comparator): usual care according to local practice
  Interventions: Other: usual care

INTERVENTIONS:
Other: usual care — Patients in the "usual care group" will be followed up according to the local practice until the end of the study.
  Arms: usual care group
Other: guideline-directed medical therapy — Patients are followed via an App, data will be evaluated by the Telemedicine team, and participants will be contacted via phone 1 week after discharge and subsequently every 7-10 days to discuss the up-titration of the HF medications.
  Other Names: telemedicine
  Arms: telemedicine guided care group

SUMMARY:
This study aims to assess the safety and effectiveness of telemedicine guided strategy on guideline-directed medical therapy (GDMT) optimization in hospitalized patients with heart failure in comparison to usual care in Switzerland.

DETAILED DESCRIPTION:
Heart failure (HF) is a chronic condition affecting approximately 26 million people worldwide, with acute decompensations leading to frequent hospitalizations and increased mortality. While guideline-directed medical therapy (GDMT) has been shown to improve outcomes in HF with reduced ejection fraction (HFrEF), real-world data indicate suboptimal implementation, with delayed initiation and low adherence to target doses. The STRONG-HF study demonstrated that rapid up-titration of GDMT following hospitalization significantly reduces HF-related mortality and readmission, highlighting the importance of early and structured treatment optimization. However, close monitoring during the vulnerable post-discharge phase remains resource-intensive and difficult to implement in routine care.

The DIGNITY study aims to assess the safety and effectiveness of a telemedicine-guided strategy for optimizing GDMT in patients with HFrEF compared to usual care in Switzerland after discharge. The study hypothesizes that telemedicine-supported management will improve GDMT optimization and clinical outcomes in this high-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at the time of hospital admission
2. Ability to use a (smart)phone and/or tablet for the follow-up
3. Documented left ventricular ejection fraction (LVEF) > 40% assessed within preceding 12 months
4. Not treated with optimal doses of oral HF therapies within 2 days before anticipated hospital discharge for acute HF in at least one of the medication categories (for details see Table 1 on page 10)
5. Hospitalized due to acute HF decompensation.
6. Specific measures within 24 hours prior to randomization

   * Systolic blood pressure > 100 mmHg, and heart rate > 60bpm
   * Serum potassium < 5mmol/L

Exclusion Criteria:

1. Inability to use a (smart)phone or tablet
2. Clear intolerance to high doses of betablockers, ACE inhibitors, or ARBs
3. Estimated glomerular filtration rate <30ml/min/1.73m2 or dialysis
4. Myocardial infarction, unstable angina or cardiac surgery within 3 months, percutaneous transluminal coronary intervention within 1 months prior to screening
5. Cardiac resynchronization therapy device implantation within 3 months prior to screening
6. Presence of significant obstructive lesion of the left ventricular outflow tract
7. Amyloid cardiomyopathy
8. Participation in other clinical trials for drugs
9. Pregnant or nursing women
10. Women of child-bearing potential who are unwilling to abstain from sexual intercourse with men or practice appropriate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
composite guideline-directed medical therapy optimization score | 3 month post-discharge
  composite guideline-directed medical therapy (GDMT) score is defined as the sum of care optimization changes and care deoptimization changes at 3 months post discharge.

SECONDARY OUTCOMES:
Proportion of clinical encounters setting 1 | during whole study phase from randomization to 90 days post-discharge
  Proportion of clinical encounters with GDMT initiations when these therapies were not used at discharge
Proportion of clinical encounters setting 2 | during whole study phase from randomization to 90 days post-discharge
  Proportion of clinical encounters with either GDMT initiations and/ or dose uptitrations, net GDMT intensification and changes in the prescription of individual GDMT elements from time to hospital admission to discharge
Dosage of diuretics | during whole study phase from randomization to 90 days post-discharge
  Requirement for decreasing or increasing dose of diuretics
Proportion of safety issues | during whole study phase from randomization to 90 days post-discharge
  Safety outcomes including incidence of hypotension, hyperkalemia, acute kidney failure (doubling of baseline serum creatinine)
Proportion of heart failure | during whole study phase from randomization to 90 days post-discharge
  Re-hospitalization due to heart failure decompensation
Proportion of hospitalization | during whole study phase from randomization to 90 days post-discharge
  All-cause re-hospitalization
Quality of life score | at randomization and 90 days post-discharge
  Quality of life (Kansas City Cardiomyopathy Questionnaire (KCCQ).
Optimization score | at randomization and 90 days post-discharge
  Optimization score is defined as the sum of care optimization changes and care deoptimization changes.
Patient Health Questionnaire | at randomization and 90 days post-discharge
  The Patient Health Questionnaire (PHQ-2) measures the frequency of depressed mood, with a score ranging from 0 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zhou, Prof. MD, Principal Investigator — Universitätsspital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided